CLINICAL TRIAL: NCT01623778
Title: Observation Study of Different Optimized Therapy Method of Patients With Chronic Hepatitis B
Brief Title: Optimization of Antiviral Therapy of Chronic HBV Infection
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, LiangXS, Assistant Professor, Changhai Hospital
Other Study IDs: HBV2012
Record Dates: First submitted 2012-06-16; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Australia Antigen Positive; Hepatitis B; Adverse Effects
Keywords: HBeAg seroconversion; Peginterferon alfa-2a; chronic hepatitis B(CHB; Optimal therapy; Response guild treatment(RGT);
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were retented at 12w,24w and 48w after optimized therapy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Add on ADV: Patients with inadequate response to interferon at 24 weeks received interferon add on ADV optimized therapy
  Interventions: Drug: Interferon Alfa-2a add on ADV
- Switch to LDT: Patients with inadequate response to interferon at 24 weeks received switching to LDT therapy
  Interventions: Drug: Interferon Alfa-2a add on ADV

INTERVENTIONS:
Drug: Interferon Alfa-2a add on ADV — Interferon add on ADV for 48 weeks
  Other Names: Response guild treatment; optimized therapy; Chronic HBV infection

SUMMARY:
Along with the improvement of the accuracy of detection of HBV serological markers, the optimization of antiviral therapy for patients with chronic hepatitis B (CHB) infection becomes feasible. Currently, the recommendation of optimized treatment especially interferon therapy are mainly based on retrospective studies, it still lacks prospective evidence. This study is aimed to evaluate the efficacy, safety and pharmacoeconomics benefits of 48 weeks optimized interferon therapy (switch to telbivudine or plus adefovir dipivoxil) for HBeAg positive CHB with inadequate response to 24 weeks interferon treatment.

DETAILED DESCRIPTION:
Patients with inadequate response to interferon therapy at 24 weeks were enrolled in this study and accepted the optimized therapy (add on ADV or switch to LDT) for 48weeks. All these patients were followed for 48 weeks and the HBeAg seroconversion and HBV DNA level were observed. Safety and the economic effect of the two optimized therapy methods also were observed.

ELIGIBILITY:
Inclusion Criteria:

patients receiving Peg interferon α-2a with inadequate response at 24 weeks (HBeAg titer ≥ 100Paul Ehrlich Institute Unit (PEIU)/ml and HBV DNA ≥ 5.0 Log copies/ml or HBV DNA titer decline <1 Log copies/ml) were enrolled into this study.

Exclusion Criteria:

* no decompensated cirrhosis,
* no hepatitis C, hepatitis D or human immunodeficiency virus (HIV) co-infection,
* no hepatocellular carcinoma and other tumors or history of severe hepatitis,
* no other systems diseases, such as a history of cardiopulmonary diseases, thyroid disorders, immune system disorders, epilepsy or mental illness (such as severe depression).

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cases of HBeAg-positive CHB with inadequate response to 24 weeks Peg interferon alpha-2a were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
HBeAg seroconversion rate | 48weeks

SECONDARY OUTCOMES:
HBV DNA decline | 48weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wan Mo Bin, Dr, Study Director — Changhai Hospital affiliated to the Second Military Medical University
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China